CLINICAL TRIAL: NCT01297283
Title: Leadless ECG Evaluation Study - Prospectively, Randomized, Cross-over, Multi-center, Interventional, Post-market Release Study to Evaluate the LECG System.
Brief Title: Leadless Electrocardiogram (ECG) Evaluation Study
Acronym: LECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Leadless ECG Evaluation Study
Record Dates: First submitted 2011-02-03; First posted 2011-02-16 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac resynchronization; Leadless ECG; Follow-up
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leadless ECG first (Experimental): Measurement of pacing thresholds are done first with the support of a leadless ECG provided by the implanted device
  Interventions: Other: LECG first
- Programmer ECG first (Active Comparator): Measurements of pacing thresholds are done first with the support of the programmer ECG
  Interventions: Other: Programmer ECG first

INTERVENTIONS:
Other: LECG first — Measurement of the pacing threshold with the support of a leadless ECG
  Arms: Leadless ECG first
Other: Programmer ECG first — Pacing threshold measurements are done with the support of the programmer ECG
  Arms: Programmer ECG first

SUMMARY:
The leadless electrocardiogram (LECG) is a new technology incorporated into the Consulta CRT-P to obtain an ECG signal from the Consulta CRT-P similar to a surface ECG obtained from the device programmer (PECG) or an external ECG machine.

The purpose of the study is to obtain more data on leadless ECG to determine whether LECG during standard CRT follow-up can indeed adequately replace surface ECG and to evaluate if it can be used during remote follow-up evaluations.

DETAILED DESCRIPTION:
The leadless electrocardiogram (LECG) is a new technology incorporated into the Consulta CRT-P to obtain an ECG signal from the Consulta CRT-P similar to a surface ECG obtained from the device programmer (PECG) or an external ECG machine. The LECG signals are measured from three electrodes mounted on the outside of the pacemaker housing and provides an electrical far field signal of the electrical activity of the heart. The LECG provides three ECG channels as different projections of the electrical activity of the heart, similar to the surface ECG. Clinical interest of LECG is threefold. First, ECG recordings are routinely used to perform pacemaker and cardiac resynchronization systems in-office follow-up mainly to determine pacing thresholds. Connection of ECG electrodes to the patient as well as the time needed to acquire an acceptable ECG signal during routine follow-up could be saved using LECG which would make follow-up easier and less time consuming. Secondly, connecting ECG electrodes requires the patient to be present at the clinic for the follow-up. Use of LECG in conjunction with a transmitting system will allow remote patient follow-up. In that case, correct ventricular capture confirmation by the LECG is of key importance. Finally, LECG stored in device memory at the time of an arrhythmia episode occurrence, can help better classify it.

The following factors might influence the quality of the LECG and/or the axis of the LECG:

* temporal changes of the electrode tissue interface due to device pocket healing process
* changes in device position and orientation over time
* body motion
* poor LECG contact due to oversized device pocket with replacement procedure. The purpose of this study is to obtain more data on leadless ECG (LECG) to determine whether LECG during standard CRT follow-up can indeed adequately replace surface ECG and to evaluate if it can be used during remote follow-up evaluations.

ELIGIBILITY:
Inclusion Criteria:

* patient with a CRT-P indication and
* patient who has signed an informed consent form.

Exclusion Criteria:

* patient younger than 18 years and/or
* unable to complete the 1-Month Follow-up visit and/or
* legally incompetent or illiterate and therefore unable to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Françoise HIDDEN-LUCET, MD, Principal Investigator — Hôpital La Pitié Salpêtrière, Paris, France
Locations (1):
- Hôpital La Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No
No sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 patients were enrolledand were followed for at least 1 month in 25 institutions in France (max 50 patients per center). The first patient was enrolled on 16th of September 2010. The last patient was enrolled on the 13th of September 2011. The last follow-up visit took place on 5th of December 2011.
Pre-assignment Details: The point of enrollment was defined as the time before device implant at which a patient has signed and dated the Informed Consent Form. At that point, the patient needed to be followed for the duration of the study (until the 1-Month Follow-Up visit) unless a Study Exit Form was completed.
Groups:
- Overall Subjects: Measurement of pacing thresholds are done first with the support of a leadless ECG provided by the implanted device
Period: Overall Study
Arm/Group | Overall Subjects
Started | 195
Completed | 176
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Overall Subjects
Number analyzed (Participants) | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (9.83)
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 80 [74 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 145
BMC Index [Mean (Standard Deviation); unit: kg/m²] | 25.64 (4.38)
Weight [Mean (Standard Deviation); unit: Kilogramms] | 72.9 (14.37)
Weight [Median (Inter-Quartile Range); unit: Kilogramms] | 71 [63 to 81]
Height [Mean (Standard Deviation); unit: meters] | 1.68 (0.09)
Height [Median (Inter-Quartile Range); unit: meters] | 1.69 [1.62 to 1.75]
BMC Index [Median (Inter-Quartile Range); unit: kg/m²] | 24.75 [22.64 to 27.76]
NYHA Class [Number; unit: participants]
  Class I | 6
  Class II | 41
  Class III | 105
  Class IV | 12
  Not available | 31
LVEF [Mean (Standard Deviation); unit: %] | 31.67 (8.18)
LVEF [Median (Inter-Quartile Range); unit: %] | 31 [25 to 35]
General cardiovascular history [Number; unit: participants]
  Cardiomyopathy | 187
  Congenital Heart Disease | 2
  Congestive Heart Failure | 29
  Coronary artery disease | 24
  Hypertension | 66
  Myocardial infarction | 25
  Pulmonary hypertension (PH) | 2
  Valve dysfunction | 26
  Other cardiovascular history | 17
Cardiovascular Surgical History [Number; unit: participants]
  NONE | 65
  Ablation | 16
  Coronary artery bypass graft (CABG) | 11
  Coronary artery intervention | 43
  Valve surgery | 20
  Other cardiovascular surgery | 5
Previous Device [Number; unit: participants]
  CRT-D implant | 6
  CRT-P implant | 39
  ICD implant | 1
  IPG implant | 37
  other | 5
Atrial Arrhythmia History [Number; unit: participants]
  NONE | 86
  Atrial fibrillation | 99
  Atrial flutter | 12
  Atrial tachycardia | 1
  Premature atrial complexes | 1
  Sinus node dysfunction | 6
  Supraventricular tachycardia | 1
  Other atrial arrhythmias | 3
Ventricular Arrhythmia History [Number; unit: participants]
  NONE | 174
  Premature ventricular complexes | 7
  Torsades de pointes | 1
  Ventricular asystole | 1
  Ventricular flutter | 1
  Ventricular tachycardia, non-sustained | 6
  Ventricular tachycardia, sustained monomorphic | 1
  Ventricular tachycardia, sustained, unknown morpho | 2
  Other ventricular arrhythmias | 3
AV Junctional Arrhythmia History [Number; unit: participants]
  NONE | 44
  1st degree AV block | 31
  2nd degree AV block | 10
  3rd degree AV block | 43
  Intermediate bundle branch block | 4
  Left bundle branch block | 96
  Right bundle branch block | 15
  Other AV junctional arrhythmias and blocks | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With LECG Performing Clinically Equivalent to PECG During Standard Pacemaker Follow-up Procedure.
Description: During CRT-P standard follow-up, ECG is used to determine atrial, left and right ventricular pacing thresholds. As primary endpoint, we will consider the proportion of patients for which for all leads LECG provides pacing threshold values that are clinically equivalent to those obtained with PECG taken as reference. The analysis will be performed on data collected at the 1-Month Follow-Up visit when the device pocket healing process is completed. Clinical equivalence will be defined as the LECG threshold values being no more than 0.5 volts different from the PECG threshold values.
Time Frame: 30 to 120 days
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Overall Subjects
Number analyzed (Participants) | 176
proportion
  Atrial lead | 0.99 (0.41) [0.95 to 1.00]
  RV Lead | 0.98 (0.56) [0.95 to 1.00]
  LV Lead | 0.98 (1.19) [0.95 to 1.00]
  All leads | 0.96 [0.92 to 0.98]

2. Secondary Outcome: Evaluation of the Possibility to Determine Ventricle Capture by an Independent Reviewer.
Description: The investigator will simulate loss of capture (LOC) at 1-Month Follow-Up visit by printing strips of LOC in both ventricular leads, LOC in LV lead only, LOC in RV lead only, no LOC. One strip randomly selected among them by the study manager will be submitted to an independent reviewer. With help of the PHD template LECG strips (intrinsic, RV paced, LV paced, BiV paced) of this patient, he/she will determine which lead is capturing.
  The endpoint is the proportion of correct classifications of ventricular capture done by then independent reviewer of LECG.
Time Frame: 30 to 120 days
Population: Proportion of Patients Correctly Classified
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Overall Subjects
Number analyzed (Participants) | 176
proportion | 0.51 [0.43 to 0.59]

3. Secondary Outcome: Evaluation of the Stability of LECG Performance Over Time.
Description: Two parameters will be used to evaluate LECG changes between PHD and 1-Month on the same LECG vector: intrinsic R wave amplitude and P waves visibility (selection the LECG vector at PHD with best combination of the highest R wave and most visible P wave).
  R wave amplitude measurements as well as P wave visibility assessment will be done by the independent reviewer.
  The endpoints evaluated are:
  * mean R wave changes from PHD to 1-month
  * proportion of patients with stable P wave visibility at PHD and 1-Month (meaning both visits visible or both visits not visible).
Time Frame: 30 to 120 days
Reporting Status: Not Posted

4. Secondary Outcome: Quality of LECG in New Devices Versus Device Replacements.
Description: The two following parameters will be used to compare the quality of LECG in new implants versus device replacements at PHD and 1-Month on the same LECG vector:
  * Intrinsic R wave amplitude
  * P waves visibility The LECG vector at PHD with best combination of the highest R wave and most visible P wave will be selected.
  R wave amplitude measurements as well as P wave visibility assessment will be done by the independent reviewer.
  The endpoints will be:
  * comparison of mean R wave values at PHD and 1-month
  * comparison of proportion of patients with P wave visible at PHD and 1-month.
Time Frame: 30 to 120 days
Reporting Status: Not Posted

5. Secondary Outcome: Effect of Posture Changes and Artifact-inducing Maneuvers on the LECG Quality.
Description: The intrinsic R wave amplitude and P waves visibility will be taken to evaluate the effect of posture changes and artifact-inducing maneuvers on the quality of LECG at the 1-Month Follow-Up visit (LECG vector with best combination of the highest R wave and most visible P wave).
  The endpoints will be R wave amplitude and P wave visibility in different positions (meaning visible or not visible in both positions).
  R wave changes and proportion of patients with stable P waves visibility at lying position versus other positions will be calculated by an independent reviewer.
Time Frame: 30 to 120 days
Reporting Status: Not Posted

6. Secondary Outcome: Evaluation of Factors Such as Device Rotation, Device Fixation, Device Side Facing the Skin, Position of Lead Loops in the Pocket, Use of Antiseptic Solution, Skin Type, Body Mass Index on the Quality of Leadless ECG.
Description: The following factors will be evaluated to investigate whether they influence the LECG quality:
  * device position (subcutaneous, submuscular, etc)
  * device rotation
  * device fixation
  * device side facing the skin
  * position of lead loops in the pocket
  * use of antibiotics in the pocket
  * skin type (loose, normal, firm)
  * body mass index (BMI)
  The endpoints will be:
  * describe R wave amplitude values
  * describe proportion of patients with P wave visible on intrinsic LECG strips recorded at 1-Month FU.
Time Frame: 30 to 120 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Overall Subjects
Serious Adverse Events (participants affected / at risk) | 35/195
Other Adverse Events (participants affected / at risk) | 3/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Subjects (N=195)
Cardiac decompensation / Global heart failure (Cardiac disorders) | 6 (8)
Phrenic nerve stimulation (Cardiac disorders) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 3 (3)
cardiogenic shock (Cardiac disorders) | 3 (3)
AV node / His ablation (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
LV lead dislodgement (Cardiac disorders) | 1 (1)
LV lead threshold elevation (Cardiac disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
Pocket hematoma (Skin and subcutaneous tissue disorders) | 4 (4)
eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Abdnominal aortic aneurysm (Vascular disorders) | 1 (1)
hepatocellular failure (Hepatobiliary disorders) | 1 (1)
allergy to iodine (Blood and lymphatic system disorders) | 1 (1)
hyperthyroidism (Endocrine disorders) | 1 (1)
fever (General disorders) | 1 (1)
multiviceral failure and cancer (General disorders) | 1 (1)
general fatigue sensation and feet formications (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Subjects (N=195)
coronary sinus dissection (Cardiac disorders) | 1 (1)
Slight deglobulisation (Blood and lymphatic system disorders) | 1 (1)
colonic ischemia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No